CLINICAL TRIAL: NCT02981784
Title: Overall Survival With Ponatinib Versus Allogeneic Stem Cell Transplant in Philadelphia-positive Leukemias With the T315I Mutation
Brief Title: Comparative Evaluation of Results of Allogeneic Hematopoietic Stem Cells Versus Ponatinib in CML Patients Carrying a Mutation T315I
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0716
Record Dates: First submitted 2016-11-21; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Leukemia
Keywords: chronic myeloid leukemia (CML); Philadelphia-positive (Ph+); Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ponatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ponatinib (PACE trial): PACE trial : "Ponatinib for Chronic Myeloid Leukemia (CML) Evaluation and Ph+ Acute Lymphoblastic Leukemia (ALL)", NCT01207440
  Interventions: Drug: Ponatinib (Iclusig®)
- Allogenis stem cell transplantation (EBMT registry): EBMT : European Group for Blood and Marrow Transplantation
  Interventions: Procedure: allogeneic stem cell transplantation

INTERVENTIONS:
Drug: Ponatinib (Iclusig®) — Novel tyrosine kinase inhibitor active in patients with an ABL T315I mutation compared to conventional or reduced intensity allogeneic stem cell transplantation.
  Groups: Ponatinib (PACE trial)
Procedure: allogeneic stem cell transplantation
  Groups: Allogenis stem cell transplantation (EBMT registry)

SUMMARY:
Effective treatment options for chronic myeloid leukemia (CML) or Philadelphia-positive (Ph+) acute lymphoblastic leukemia (ALL) patients with the T315I mutation are few. This study compared overall survival (OS) between CML and Ph+ ALL patients treated with ponatinib versus allogeneic stem cell transplantation (allo-SCT).

ELIGIBILITY:
Inclusion Criteria:

* CML any phase with T315I mutation
* Ph+ ALL with a T315I mutation
* Being treated in the PACE trial according to the criteria of this phase II trial
* Or being allogeneic stem cell transplanted with any source of allogeneic cells and after any conditioning regimen.

Exclusion Criteria:

* Ph negative patients
* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All 128 T315I+ patients from PACE comprised the ponatinib group of this study. Fifty-six patients from the EBMT database comprised the allo-SCT group
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2000-01; Primary Completion 2011-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival after either allogeneic stem cell transplantation or Ponatinib initiation. (Time between therapeutic intervention and death, in months) | From date of inclusion until the date of death, assessed up to 180 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon-Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No